CLINICAL TRIAL: NCT05113784
Title: A Multicenter, Double-blind, Randomized Controlled, add-on Phase 2/3 Study of the Safety and Efficacy of Meplazumab in Patients With COVID-19
Brief Title: the Safety and Efficacy of Meplazumab in Patients With COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPZ-II-01-CN
Record Dates: First submitted 2021-09-17; First posted 2021-11-09 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — meplazumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meplazumab for Injection (Experimental): First dose: 0.2 mg/kg - Day 1; Second dose: 0.2 mg/kg - Day 8
  Interventions: Drug: Meplazumab for Injection
- Placebo (Placebo Comparator): First dose: control - Day 1; Second dose: control -Day 8
  Interventions: Drug: Sterile normal saline (0.9%)

INTERVENTIONS:
Drug: Meplazumab for Injection — humanized antibody target CD147
  Arms: Meplazumab for Injection
Drug: Sterile normal saline (0.9%) — Sterile normal saline (0.9%)
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled phase 2/3 clinical study. Based on the results of the Phase I clinical study, one repeat dose group and one placebo group are used for the standard treatment of the Novel Coronavirus Pneumonia Protocol (Trial 8) The treatment regimen is a one-time intravenous infusion of either mprozumab or placebo on day 1 (D1) and day 8 (D8) of the treatment period at a dose of 0.2 mg/kg based on body weight. An estimated 150 subjects will be randomly assigned to either Meplazumab or placebo in a 2:1 ratio A short-term efficacy evaluation was performed to determine the efficacy and safety of Meplazumab in each subject within 14 days of initial administration and a long-term follow-up evaluation was performed 28 days after initial administration to determine the safety of Meplazumab.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤Subject ≤ 75 years, Male and/or female;
* Clinical confirmation of COVID-19 patients in accordance with novel Coronavirus Diagnosis and Treatment Protocol (Trial Version 8) of the NHC
* Participants must be able to understand and willing to participate in this research, this study and signed informed consent form (if incapacitated subjects, the researchers believe the subjects to the test in its own interests, should be signed by its legal guardian informed consent, or telephone inform consent (recording) and note it in the original medical records and other relevant documents)

Exclusion Criteria:

* Subjects with any unstable conditions, a history of significant hypersensitivity, or known allergy to components of the investigational agent;
* SARS-CoV-2 infection by PCR ≥ 96h;
* Platelet (PLT) < 50×10^9/L, or hemoglobin (HGB) < 60g/L;
* Total bilirubin (TBIL) > 2×ULN (upper limit of normal value), or alanine transferase (ALT), aspartate transferase (AST), alkaline phosphatase (ALP) > 5×ULN;
* glomerular filtration rate (GFR) < 30mL/min·1.73m^2, or serum creatinine increased by 0.5mg/ dL within 7 days, or oliguria (<400mL/24hr), or anuria (<100mL/24hr);
* Pregnant or breast feeding;
* Persons who have family planning or do not agree to use effective non-drug contraceptive measures within 6 months after signing the ICF;
* Subjects participating in another clinical study. There will be a need for washout with 5 half lives depending on the study treatment or 30 days since any previous study, whichever is longer;
* he inestigators concluded that the patients had other reasons for not being eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Time of virus nucleic acid test turning negative | up to 14 days
  Time of virus nucleic acid test turning negative

SECONDARY OUTCOMES:
Treatment to discharge time | up to 28 days
  Treatment to discharge time
Evolution of the imaging parameters | up to day28
  Changes from pre-dose baseline in CT
Assessment of the immune response profile | up to day28
  Immune response profile characterized according immune cells and subsets and CRP.
Assessment of the biochemistry profile | up to day28
  Change from pre-dose baseline in blood biochemistry:Fbg,Cr,BUN,UA,AST,ALT,g-GT,TBIL,ALB,TP,NA,K,Ca,CL
Assessment of the cytokines profile | up to day28
  Change from pre-dose baseline in cytokines:IL-1b、IL-6、IL-8、IL-10、IL-17、CCL2、CXCL-1、CXCL-2、IFN-γ、TNFα、CyPA

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Principal Investigator — Shenzhen Third People's Hospital; Yinzhong Shen, Principal Investigator — Shanghai Public Health Clinical Center; Yingxia Liu, Principal Investigator — Shenzhen Third People's Hospital
Locations (2):
- China (2):
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The Third People's Hospital Of Shenzhen, Shenzhen